CLINICAL TRIAL: NCT05047055
Title: Multi-centric Prospective Cohort Study of TB Recurrence Free Cure Among Microbiologically Confirmed New Pulmonary Tuberculosis Patients Treated Under NTEP With the 4-month Moxifloxacin Containing Daily Regimen
Brief Title: Four Months Moxifloxacin Containing Daily Regimen Study Among New Pulmonary Tuberculosis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: Indira Gandhi Government Medical College and Hospital (IGGMCH), Nagpur (Unknown); King George's Medical University, Lucknow (Unknown); Mahavir Hospital and Research Centre, Hyderabad (Unknown); Government Vellore Medical College and Hospital, Adukkamparai (Unknown); Lok Nayak hospital, New Delhi (Unknown)
Responsible Party: Principal Investigator, Banu Rekha, Scientist E, Tuberculosis Research Centre, India
Other Study IDs: 2021010
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid; Protons; Rifampin; Pyrazinamide; Ethambutol; Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum sample of Mycobacterium Tuberculosis with its DNA will be preserved (Positive sputum isolates at baseline and at the time of TB recurrence will be sent to ICMR-NIRT, Chennai for storage for future genotyping)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group - 4 months moxifloxacin group: Isoniazid (H), Rifampicin (R), Pyrazinamide (Z), Ethambutol (E), Moxifloxacin (M)
  Isoniazid, rifampicin, pyrazinamide, ethambutol and moxifloxacin daily for 2 months followed by isoniazid, rifampicin, ethambutol and moxifloxacin daily for 2 months (2 HRZEM daily / 2HREM daily) - Duration 4 months
  Drug dosages The Fixed-dose Combination (FDC) for HRZE(75/150/400/275mg) used under NTEP according to weight category will be used.
  The patients enrolled in the study will receive an additional tablet of moxifloxacin(M) 400mg (body weight <64 Kg) / 600mg (body weight >65 Kg) along with the FDC both in the intensive and continuation phase.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Isoniazid — Intensive Phase for 2 months and Continuation phase for 2 months dose: 75 mg (2 tablets for 30 - 34 Kg, 3 tablets for 35 - 49 Kg, 4 tablets for 50 - 64 Kg, 5 tablets for 65 - 75 Kg and 6 tablets for >75 Kg) as a fixed-dose combination.
  Other Names: H
Drug: Rifampicin — Intensive Phase for 2 months and Continuation phase for 2 months dose: 150 mg (2 tablets for 30 - 34 Kg, 3 tablets for 35 - 49 Kg, 4 tablets for 50 - 64 Kg, 5 tablets for 65 - 75 Kg and 6 tablets for >75 Kg) as a fixed-dose combination.
  Other Names: R
Drug: Pyrazinamide — Intensive Phase for 2 months only dose: 400 mg (2 tablets for 30 - 34 Kg, 3 tablets for 35 - 49 Kg, 4 tablets for 50 - 64 Kg, 5 tablets for 65 - 75 Kg and 6 tablets for >75 Kg) as a fixed-dose combination.
  Other Names: Z
Drug: Ethambutol — Intensive Phase for 2 months and Continuation phase for 2 months dose: 275 mg (2 tablets for 30 - 34 Kg, 3 tablets for 35 - 49 Kg, 4 tablets for 50 - 64 Kg, 5 tablets for 65 - 75 Kg and 6 tablets for >75 Kg) as a fixed-dose combination.
  Other Names: E
Drug: Moxifloxacin — Intensive Phase for 2 months and Continuation phase for 2 months dose: 400 mg for 30 to 64 yrs AND 600 mg for 65 and above years of age.
  Other Names: M

SUMMARY:
The 4-month daily regimen containing moxifloxacin (2HRZEM 7 / 2HRM7) of ICMR-NIRT was studied in 321 sputum positive pulmonary TB patients in a randomised clinical trial. Of the 321, there were 96% with sputum smear grading of 2+/3+ and 80% with >2 zone involvement in the chest radiograph, The sputum culture conversion at the end of intensive phase was 94%, favourable response at the end of treatment of 92% and the TB recurrence rate was 4.1%. The regimen was safe and well tolerated.

The advantages of a 33% reduction in treatment duration are manifold in terms of financial and other administrative implications. As the next logical step investigators believe that the effectiveness of this shortened regimen that proved successful in our study needs to be tested in the field. Under NTEP the anti-TB drugs are offered as Fixed dose Combination (FDC).3 The HREZ intensive phase and HRE continuation phase FDC are administered to patients based on body weight category. If our proposed study proves successful, the addition of moxifloxacin tablet to the FDC of anti-TB drugs in the intensive and continuation phases of treatment would be feasible under TB program settings. Investigators propose to evaluate 4-month moxifloxacin containing daily regimen [2 months of HRZEM daily / 2 months of HREM daily (2 HRZEM 7 / 2HREM7)] in the treatment of newly diagnosed sputum smear positive pulmonary TB patients.

DETAILED DESCRIPTION:
Scientific rationale The 4-month daily regimen containing moxifloxacin (2HRZEM 7 / 2HRM7) of ICMR-NIRT was studied in 321 sputum positive pulmonary TB patients in a randomised clinical trial.7 Of the 321, there were 96% with sputum smear grading of 2+/3+ and 80% with >2 zone involvement in the chest radiograph, The sputum culture conversion at the end of intensive phase was 94%, favourable response at the end of treatment of 92% and the TB recurrence rate was 4.1%. The regimen was safe and well tolerated.

The advantages of a 33% reduction in treatment duration are manifold in terms of financial and other administrative implications. As the next logical step investigators believe that the effectiveness of this shortened regimen that proved successful in our study needs to be tested in the field. Under NTEP the anti-TB drugs are offered as Fixed dose Combination (FDC). The HREZ intensive phase and HRE continuation phase FDC are administered to patients based on body weight category. If our proposed study proves successful, the addition of moxifloxacin tablet to the FDC of anti-TB drugs in the intensive and continuation phases of treatment would be feasible under TB program settings. Investigators propose to evaluate 4-month moxifloxacin containing daily regimen [2 months of HRZEM daily / 2 months of HREM daily (2 HRZEM 7 / 2HREM7)] in the treatment of newly diagnosed sputum smear positive pulmonary TB patients.

Objectives :

Primary objective:

To determine the TB recurrence free cure rate among microbiologically confirmed new pulmonary tuberculosis (PTB) patients treated under NTEP with the 4-month moxifloxacin containing daily regimen.

Secondary objectives:

1. To determine the Adverse drug reactions (ADR) with the 4-month moxifloxacin containing daily regimen
2. To determine to response to treatment with the 4-month moxifloxacin containing daily regimen
3. To store paired samples of culture isolates of patients with TB recurrence for future genotyping.

Study sites: Nagpur, Lucknow, Delhi, Hyderabad, Vellore (5 sites) Study population: Newly diagnosed adult sputum smear and or CBNAAT positive PTB patients

Sample size calculated was 550 patients.

Screening assessments Clinical evaluation, Laboratory evaluations will be done initially.

Positive sputum isolates at baseline and at the time of TB recurrence will be sent to ICMR-NIRT, Chennai for storage for future genotyping.

Follow-up Follow-up during treatment: During the treatment phase the patients will be followed every month

Follow-up post- treatment :

During post-treatment, the patients will be followed up once in 3 months at 3, 6, 9 and 12 months and once every six months upto 24 months (ie. at 18 and 24 months). The 95% confidence interval of the TB recurrence free cure rate will be used to conclude on the performance of the 4 month moxifloxacin containing regimen under program settings.

Study duration:

Recruitment, training of staff: 2 month Duration of enrollment : 10 months Duration of treatment: 4 months Follow-up period : 24 months post-treatment Data analysis and report generation : 2 months Total study duration: 3.5 years

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. At least one sputum smear and or CBNAAT test should be positive for tubercle bacilli
3. Female participants of childbearing potential must have a negative urine pregnancy test at screening. Those who have not undergone permanent sterilisation - tubal ligation or spouse with vasectomy must agree for use of contraceptive measures for birth control - vaginal diaphragm, intrauterine device, condom until treatment completion.
4. Willing to follow the trial procedures
5. Willing to give written informed consent
6. Residing within the study TU

Exclusion Criteria:

1. Body weight less than 30 kg
2. Previous anti-TB treatment, if any, should not exceed one month in the past 2 years and more than 7 days in the preceding one month
3. Multidrug resistant TB (MDR-TB)
4. Resistance to isoniazid or rifampicin or quinolone as evidenced by Cartridge based Nucleic acid Amplification test (CBNAAT) and Line probe Assay (LPA) test
5. Associated extra-pulmonary TB except TB superficial lymphadenitis
6. Hepatic or renal disease as evidenced by clinical or biochemical abnormalities- ALT/AST> 2.5 times ULN or Total bilirubin >1.2 mg/dl, Serum Creatinine >1.2 mg/dl, Blood Urea >43 mg/dl.
7. QTcF> 450 ms or bundle branch block or heart block on ECG
8. Psychiatric illness
9. Seizure disorder
10. Pregnancy or lactation
11. Those seriously ill as defined by a score of <50 on Karnofsky scale (Annexure 1)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed adult sputum smear and or CBNAAT positive pulmonary TB patients
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
TB recurrence free cure | 24 months after treatment
  The proportion of microbiologically confirmed new PTB patients with TB recurrence free cure among those treated with the 4-month moxifloxacin containing daily regimen.

SECONDARY OUTCOMES:
Adverse drug reaction | 4 months, at the end of treatment
  The proportion of PTB patients with adverse drug reactions in those treated with the 4-month moxifloxacin containing daily regimen.
TB Sustained treatment Success, failure, death, loss to follow up | 10 months
  The proportion of PTB patients with sustained treatment success, failure, death, lost to follow-up
TB Relapse and Reinfection | 24 months after treatment
  The proportion of patients with TB relapse and TB re-infection based on genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Banurekha MBBS., MPH, Principal Investigator — National Institute for Research in Tuberculosis, Chennai, India
Locations (1):
- National Institute for Research in Tuberculosis, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No